CLINICAL TRIAL: NCT06698705
Title: Electroencephalogram Study in Children Under Remimazolam Anesthesia - a Prospective,Observational Study
Brief Title: The EEG Study Under Remimazolam Anesthesia in Children
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2024-03-221
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Electroencephalography; Remimazolam; Child Neglect
Keywords: Electroencephalography; Remimazolam; children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1-3 years: The child should wear EEG consumables accompanied by their family and be properly secured in the operating room. Induction and maintenance of Remimazolam, collection of EEG information . EEG collection covers the entire perioperative period, including preoperative awake period (or preoperative sedation period), surgical anesthesia period, and anesthesia awake period.
- 4-6 years: The child should wear EEG consumables accompanied by their family and be properly secured in the operating room. Induction and maintenance of Remimazolam, collection of EEG information . EEG collection covers the entire perioperative period, including preoperative awake period (or preoperative sedation period), surgical anesthesia period, and anesthesia awake period.
- 7-12 years: The child should wear EEG consumables accompanied by their family and be properly secured in the operating room. Induction and maintenance of Remimazolam, collection of EEG information . EEG collection covers the entire perioperative period, including preoperative awake period (or preoperative sedation period), surgical anesthesia period, and anesthesia awake period.

SUMMARY:
The effect of Remimazolam on brain electrical activity. Previous studies have shown that in healthy male volunteers, EEG changes during Remimazolam infusion are characterized by an initial increase in the beta band and a later increase in the delta band. When monitoring the depth of anesthesia, the commonly used Bispectral Index in clinical practice was originally developed for propofol. Therefore, studies have shown that the correlation between the depth of sedation of benzodiazepines such as midazolam and Bispectral Index is weak. In contrast, the beta wave ratio is considered a more suitable EEG indicator for monitoring the sedative effect of Remimazolam. The above indicates that Remimazolam has a specific pattern of influence on EEG activity, especially in the regulation of anesthesia depth, with unique characteristics.

DETAILED DESCRIPTION:
This study is a prospective, observational study.Children undergoing elective general anesthesia with Remimazolam will be divided into three groups (1-3 years old, 4-6 years old, 7-12 years old) based on their age range, with 20 cases in each group.Inform the family of the general research plan and obtain informed consent. Main outcome measure: Time frequency characteristics of electroencephalography (EEG) in children of different age groups under general anesthesia withRemimazolam (including anesthesia induction, maintenance, and recovery periods).

ELIGIBILITY:
Inclusion Criteria:

1. aged 1 years-12 years; 2, with American Society of Anesthesiologists (ASA) physical status I or II; 3, children requiring general anesthesia under remimazolam; 4, parents or legal guardians of children who volunteered to participate in the trial; And signed the informed consent form.

Exclusion Criteria:

1. Congenital malformation or other genetic conditions that are thought to affect brain development ;
2. History of severe heart, brain, liver, kidney and metabolic diseases ;
3. Premature infants (≤32 weeks);
4. Upper respiratory tract infection in the last two weeks. -

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children were aged 1 years-12 years; with American Society of Anesthesiologists (ASA) physical status I or II; and requiring general anesthesia under remimazolam;
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time-frequency characteristics of electroencephalogram (EEG) | Intraoperative (during remimazolam general anesthesia (including anesthesia induction, maintenance and recovery)
  Time-frequency characteristics of electroencephalogram (EEG) in children of different ages during remimazolam general anesthesia (including anesthesia induction, maintenance and recovery) .

SECONDARY OUTCOMES:
Modified observer's assessment of alertness/sedation (MOAA/S) | Intraoperative (during remimazolam general anesthesia (including anesthesia induction, maintenance and recovery)
  5#Subject responds readily to name spoken in a normal tone; 4 #Lethargic response of a subject to a name spoken in a normal tone; 3 #The subject responds only after a name is called loudly and repeatedly; 2 #The subject responds only after mild prodding or shaking;
  1 #The subject responds only after a painful trapezius squeeze; 0 #The subject does not respond to painful trapezius squeeze. MOAA/S score ≤ 2 points represent successful sedation
Recovery time | Within up to 30 minutes after operation
  From the time sevoflurane was stopped until the child opened his eyes for the first time and reached an Aldrete score of ≥9
Pediatric anesthesia emergence delirium | Within up to 30 minutes after operation
  The pediatric anesthesia emergence delirium scale consists of four items. Each item is scored 0-4 yielding a total between 0 and 20. The degree of emergence delirium increased directly with the total score.
The Face, Legs, Activity, Cry, Consolability Scale (FLACC) | Within up to 30 minutes after operation
  The FLACC scale consists of five items. Each item is scored 0-2 yielding a total between 0 and 10. The degree of pain increased directly with the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Yuhang Cai, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China